CLINICAL TRIAL: NCT06208670
Title: The Effect of Progressive Muscle Relaxation Exercises Given to Women Experiencing Premenstrual Syndrome on Premenstrual Syndrome Symptoms and Tendency to Violence
Brief Title: Progressive Muscle Relaxation Exercises on Premenstrual Syndrome
Acronym: PMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Sabri Togluk, Lecturer Doctor, Siirt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STogluk
Record Dates: First submitted 2023-12-22; First posted 2024-01-17 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual Syndrome Symptoms; Tendency to Violence; Progressive Muscle Relaxation Exercises
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation Exercises (Experimental): Progressive Relaxation Exercises (PGE) Practice: The importance and benefits of PGE exercises, situations to be avoided during the exercise, and the process of teaching by practicing and practicing the exercise will be done by the trained researcher for eight weeks, and it will be ensured that they repeat it at home. Progressive relaxation exercise instructions and a practical demonstration of the researcher will be made with the directives in the audio video with music. During the relaxation exercises, individuals will first intentionally tighten the muscle groups in the hands, arms, neck, shoulders, face, chest, abdomen, buttocks, feet, and fingers (muscle groups starting from the hands and ending with the feet) and then relax the muscles according to the commands on the CD.
  Interventions: Behavioral: Progressive muscle relaxation exercises
- Violent tendency Scale (Experimental): was developed to identify aggression and violence tendencies
  Interventions: Behavioral: Violent tendency Scale

INTERVENTIONS:
Behavioral: Progressive muscle relaxation exercises — PMI is among the non-pharmacological methods nurses can offer caregivers (Yılmaz et al., 2019). Health professionals, especially nurses, should evaluate all women of reproductive age in terms of PMS, plan educational interventions that will increase their awareness of the issue and enable them to develop appropriate coping strategies, support the planned educational interventions through written or visual materials, provide effective and quality counseling services, and aim to improve women's decreased quality of life (Abay & Kaplan 2019; Aksoy Derya et al. 2019; Akmalı et al. 2020). Women can be advised to do relaxation exercises such as walking, running, swimming, and yoga regularly (at least 30 minutes a day) as they reduce stress by increasing endorphin levels and improve heart rate, lung capacity, and general health (Penedo & Dahn, 2005; ACOG, 2015; Khajehei 2015).
  Arms: Progressive Muscle Relaxation Exercises
Behavioral: Violent tendency Scale — Violent tendency Scale
  Arms: Violent tendency Scale

SUMMARY:
Abstract Purpose: This study was conducted to determine the effect of progressive muscle relaxation exercises given to women experiencing premenstrual syndrome on premenstrual syndrome symptoms and tendency to violence.

Materials and Methods: The research was planned as an experimental study with a pretest-posttest control group, with female patients coming for examination at Siirt Training and Research Hospital Gynecology Polyclinics between December 2023 and August 2024. "Personal Information Form, Premenstrual Syndrome Scale and Violence Tendency Scale" were used to collect data in the study. Percentage distributions and t-test in independent groups were used to evaluate the data.

DETAILED DESCRIPTION:
Premenstrual Syndrome (PMS) is defined as a set of physical, psychological, and behavioral symptoms that occur about five days before menstruation and disappear within a few days following its onset (Ryu & Kim, 2015). In a systematic study evaluating data from 17 countries, the prevalence of PMS was 47.8% (Direkvand-Moghadam et al., 2014). In a systematic study conducted to investigate the prevalence of PMS in women of reproductive age in Turkey, the overall prevalence was determined as 52.2%. It was reported that PMS was seen in 59% of high school students, 50.3% of university students, and 66% of the general female population (Erbil & Yücesoy, 2021). Although there are many different symptoms associated with PMS, common physical symptoms include abdominal bloating, weight gain, fatigue, breast tenderness, skin problems, dizziness, and headache or joint pain. Common psychological and behavioral symptoms include mood swings, anger, anxiety, aggression, sad or depressed mood, appetite changes, difficulty concentrating, and decreased interest in activities (Women's Health Concern 2012, Gunderson and Yates 2013; Yonkers & Casper, 2022c). Symptoms related to PMS are reported to cause difficulty in attending school or work, a decline in academic achievement, economic losses, deterioration in interpersonal relationships, social isolation, risk of suicide attempt, substance abuse, and increased tendency to commit crimes or accidents (Borenstein et al., 2003; Yonkers et al., 2008; Tadakawa et al. 2016; Buddhabunyakan et al. 2017, Owens and Eisenlohr-Moul 2018, Abay and Kaplan 2019, Schoep et al. 2019a, 2019b). In addition, the tendency to violence, domestic fights, and child abuse have been reported in women diagnosed with PMS (Halberich, 2007). At the cognitive level, all of the positive thoughts that a person who is ready for violence attributes to violence can be defined as violent tendencies (Karaboğa, 2018). It is known that incidents of violence are increasing in our country, especially among young people (TBMM 2007). On the other hand, violence and aggression are essential problems that are becoming increasingly common all over the world (WHO2002, WHO 2014).

The treatment of PMS is usually carried out gradually, including non-pharmacological strategies, pharmacological strategies, including antidepressants or hormonal methods, and surgery (Walsh et al., 2015). PGE, first developed by the American Dr. Jacobson in the 1920s, involves each muscle group's contraction and relaxation, respectively (Liu et al., 2020). During PGE, the major muscle groups are followed in a specific order; this order is hands, arms, eyebrows, eyes, back of neck, front of neck, shoulders, back, chest, abdomen, buttocks, front of thigh, back of thigh, calf and feet (Bushra & Ajaz, 2018; Dhyani et al., 2015; Liu et al., 2020; Perakam et al., 2019). Progressive relaxation exercise is a breathing and stretching method that provides relaxation of nerves and muscles from hand to foot, stimulating the parasympathetic nervous system and reducing sympathetic nervous system activities. In this way, blood pressure, heart and respiratory rate slow down, metabolic rate decreases, endorphin release, pain, and fatigue, and facilitate the transition to sleep (Özer & Ergen, 2010; Kurt & Kapucu, 2018).

PGE is among the non-pharmacological methods that nurses can offer caregivers (Yılmaz et al., 2019). It is necessary for health professionals, especially nurses, to evaluate all women of reproductive age in terms of PMS, to plan educational interventions that will increase their awareness of the issue and enable them to develop appropriate coping strategies, to support the planned educational interventions through written or visual materials, to provide effective and quality counseling services, and to aim to improve women's decreased quality of life (Abay & Kaplan, 2019; Aksoy Derya et al. 2019, Akmalı et al 2020). Women may be advised to do relaxation exercises such as walking, running, swimming, and yoga regularly (at least 30 minutes a day) as they reduce stress by increasing endorphin levels and improve heart rate, lung capacity, and general health (Penedo & Dahn 2005; ACOG 2015; Khajehei 2015).

The study aimed to determine the effect of progressive muscle relaxation exercises given to women with premenstrual syndrome on premenstrual syndrome symptoms and violent tendencies.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in the study,
2. 18-40 years old,
3. At least primary school graduate,
4. Scored 110 and above on the Premenstrual Syndrome Scale,
5. Menstrual cycle length for the last three months is within normal limits (21-35),
6. Women who have not used oral contraceptives for the last three months.

Exclusion Criteria:

1. Having a physical or mental illness that would prevent participation in the study,
2. Women who score below 110 points on the Premenstrual Syndrome Scale.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The reason why we included only female subjects in our study is that we studied premenstrual syndrome as a subject.
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale | Six month
  The premenstrual Syndrome Scale (PMSS) was developed by Başaran GENÇDOĞAN in 2006. The scale consists of 44 items in a 5-point Likert type (never, very rarely, sometimes, frequently, continuously). In the scoring of the scale, 1= never, 2= very rarely, 3= sometimes, 4= frequently, 5= continuously. A minimum score of 44 and a maximum score of 220 can be obtained from the scale. The reliability of the PMSQ was determined by test-retest and internal consistency methods. The reliability of the scale is Cronbach's alpha 0,75. (Gençdoğan, 2006).

SECONDARY OUTCOMES:
The Violence Tendency Scale | Six month
  The Violence Tendency Scale (VTS) was developed by Göka, Bayat, and Türkçapar (1995) to determine aggression and violence tendencies and was redesigned in the research on "Violence in the Family and the Social Sphere" (1998) conducted by the Turkish Prime Ministry Family Research Institute without changing its basic structure and content validity was ensured. The scale includes 20 questions graded between 1-4. On the scale, 1-20 points indicate (a very low tendency to violence), 21-40 points (a low tendency to violence), 41-60 points (a high tendency to violence), and 61-80 points (a very high tendency to violence) (29).

CONTACTS AND LOCATIONS:
Overall Officials: Sidar GÜL, PhD, Study Chair — SİİRT UNIVERSITY
Locations (1):
- Siirt Education Research Hospital, Siirt, Centrum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Once our study is finalized, it is planned to be published in an international journal.
Supporting Information: SAP, CSR
Time Frame: The data will be made available at the end of the study and there will be no restrictions on use.
Access Criteria: Attribution Use for scientific purposes

REFERENCES:
- [Derived] Togluk S, Gul S. The effects of progressive muscle relaxation exercises on premenstrual syndrome symptoms and violence tendencies in women: a randomized controlled trial. BMC Womens Health. 2025 Apr 12;25(1):176. doi: 10.1186/s12905-025-03712-4. PMID 40221724